CLINICAL TRIAL: NCT03022617
Title: An Investigator Initiated Open Label Study Evaluating the Efficacy and Tolerability of Oral Apremilast for the Treatment of Nail Psoriasis
Brief Title: A Study Evaluating the Efficacy and Tolerability of Oral Apremilast for the Treatment of Nail Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Boni Elewski, Professor, Chairman, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-160720004
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Psoriatic Nail; Psoriasis Vulgaris; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Open-label drug administration group. No comparator.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast

SUMMARY:
Psoriasis vulgaris is a common inflammatory condition of the skin that results in scaly red itchy plaques. In addition to affecting the skin, psoriasis can also cause disease in the finger and toe nails. The most characteristic nail findings associated with nail psoriasis are nail pitting, onycholysis with a rim of erythema, and oil spots. Because nail psoriasis causes a substantial disease burden for patients, it is critical that safe and effective treatments are found for this specific type of psoriasis. Unfortunately, nail psoriasis is often difficult to treat.

Apremilast is an orally available small molecule inhibitor of phosphodiesterase 4 (PDE4) that is FDA approved for the treatment of psoriasis and psoriatic arthritis. Apremilast has shown promising results for treating psoriatic arthritis and nail disease; however more data is needed regarding its effect on nail psoriasis (Kavanaugh, et al). We hypothesize that apremilast will prove to be highly effective in treating nail psoriasis. We propose to conduct an open label clinical trial to investigate the efficacy and tolerability of apremilast in treating nail psoriasis, where we will follow the package insert guidelines for treating patients with apremilast.

DETAILED DESCRIPTION:
Psoriasis vulgaris is a common inflammatory condition of the skin that results in scaly red itchy plaques. In addition to affecting the skin, psoriasis can also cause disease in the finger and toe nails. Nail psoriasis is a chronic disease and can present with the following clinical findings: splinter hemorrhage, leukonychia, red spots in the lunula, nail pitting, nail plate crumbling, hyperkeratosis, and/or nail plate separation from the nail bed. The most characteristic nail findings associated with nail psoriasis are nail pitting, onycholysis with a rim of erythema, and oil spots. Special interest will be paid to identifying these particular nail findings in patients, however all potential nail psoriasis symptoms will be assessed in patients in this study. Due to the highly visible nature of disease in the fingernails, nail psoriasis often results in a substantial deleterious effect on a patient's quality of life. Patients also can have significant pain and disability due to nail psoriasis.

Psoriasis patients who have nail involvement are known to have more severe psoriasis disease and diminished quality of life when compared to psoriasis patients without nail disease. Patients with nail psoriasis often also have psoriatic arthritis, and untreated psoriatic arthritis is known to lead to joint destruction with potentially severe morbidity. Nail psoriasis has a reported incidence of 80 to 90% (Jiaravuthiasan, et al). Because nail psoriasis causes a substantial disease burden for patients, it is critical that safe and effective treatments are found for this specific type of psoriasis. Unfortunately, nail psoriasis is often difficult to treat.

Apremilast is an orally available small molecule inhibitor of phosphodiesterase 4 (PDE4) that is FDA approved for the treatment of psoriasis and psoriatic arthritis. PDE4 is one of the main phosphodiesterases expressed in immune cells, and its inhibition by apremilast is thought to increase cyclic adenosine monophosphate and thereby decrease the inflammatory response. Specifically, apremilast is believed to down regulate pro-inflammatory cytokines including TNF-α, (Tumor necrosis Factor) IL-23 (Interleukin), IL-17, and others.

Apremilast has shown promising results for treating psoriatic arthritis and nail disease; however more data is needed regarding its effect on nail psoriasis (Kavanaugh, et al). We hypothesize that apremilast will prove to be highly effective in treating nail psoriasis. We propose to conduct an open label clinical trial to investigate the efficacy and tolerability of apremilast in treating nail psoriasis, where we will follow the package insert guidelines for treating patients with apremilast.

ELIGIBILITY:
Inclusion Criteria:

* - Patients older than 18
* Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
* Be willing and consent to having photos taken of their fingernails
* Diagnosis of chronic plaque psoriasis that has been present for at least 6 months prior to baseline
* Plaque psoriasis involving at least 5% of the patient's body surface area
* Nail psoriasis in at least one finger nail with a mNAPSI of 5 or greater
* A Nail Pain VAS score of 4 or higher. The Nail Pain VAS will assess the severity of pain linked to the nail disease.
* Must have discontinued all systemic therapies for the treatment of psoriasis or psoriatic arthritis at least 4 weeks or 5 half-lives, and biologics 2 months or 5 half-lives (whichever is longer) prior to baseline visit
* Must have discontinued all topical therapies for the treatment of psoriasis at least 2 weeks prior to baseline visit
* Subjects must have discontinued UV therapy at least 2 weeks prior to baseline and PUVA (psoralen ultraviolet light therapy) at least 4 weeks prior to baseline.
* Subjects must be in good general health without significant uncontrolled comorbidities, other than psoriasis, as determined by the investigator based on exam findings, medical history, and clinical laboratories. Patients with stable mild renal insufficiency are eligible for enrolling in this trial.
* Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the last dose of apremilast, and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, partners vasectomy, or male or female condoms that are not made of natural materials plus a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide. Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).
* Male subjects, including those who have had a vasectomy, must use condoms not made of natural materials for the duration of the trial and for at least 28 days after the last dose of apremilast if conception is possible.

Exclusion Criteria:

* - Unable to comply with the protocol (as defined by the Investigator; i.e. drug or alcohol abuse or history of noncompliance)
* Pregnancy or breastfeeding
* Female patients of childbearing potential and male patients who engage in activity where contraception is possible who are unable to use the approved methods of contraception throughout the length of the study and 28 days following the last dose
* Patients who have or have had thoughts of suicide or hurting themselves.
* Patients with prior exposure to apremilast
* Subject has been treated with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to baseline visit.
* Patients with severe, progressive, or uncontrolled medical or psychiatric disease.
* Concomitant therapy with medications that are strong cytochrome P450 inducers, including rifampin, phenobarbital, carbamazepine, or phenytoin
* Any other dermatologic conditions that prohibit or confound the ability of the investigator to interpret skin and/or nail exam findings.
* Patients who will be unable to avoid the use of systemic steroids, excluding intranasal or inhaled steroids that will be permitted, for the duration of the trial
* Any known hypersensitivity to apremilast
* Any subject who, in the opinion of the investigator, will be uncooperative or unable to comply with duty procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01; Primary Completion 2020-09-01 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Open-label drug administration group. No comparator.
  Apremilast
Period: Overall Study
Arm/Group | Study Group
Started | 12
Completed | 6
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change of mNAPSI (Modified Nail Area Psoriasis Severity Index) at Week 36 Compared to Baseline for All Nails.
Description: mNAPSI is an objective scoring system administered by trained health care providers. Scores range from 0 (no nail disease) to 130 (complete nail involvement in all ten nails.)
Time Frame: 36 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of reduction in mNAPSI score
Arm/Group | Study Group
Number analyzed (Participants) | 6
percentage of reduction in mNAPSI score | 64.1 [46.5 to 81.7]
Statistical Analysis 1: Comparison: Study Group; Test type: Superiority; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 21.5, Standard Deviation 10.89

2. Secondary Outcome: Mean Percent Change in mNAPSI of Target Nail at Weeks 12, 24, 36, 48, and 52 Compared to Baseline.
Description: The target nail will be defined as the nail that has the highest mNAPSI singe nail score at baseline. This nail will remain the target nail for the remainder of the study. mNAPSI is an objective scoring system administered by trained health care providers. Scores range from 0 (no nail disease) to 130 (complete nail involvement in all ten nails.)
Time Frame: 12, 24, 36, 48, and 52 weeks
Population: Participants lost to follow-up
Measure: Mean (95% Confidence Interval); unit: percentage of reduction in mNAPSI score
Arm/Group | Study Group
Number analyzed (Participants) | 11
percentage of reduction in mNAPSI score
  Week 12 | 53.9 [0 to 100]
  Week 24: number analyzed (Participants) | 9
  Week 24 | 65.1 [40 to 100]
  Week 36: number analyzed (Participants) | 6
  Week 36 | 63.8 [20 to 100]
  Week 48: number analyzed (Participants) | 6
  Week 48 | 57.7 [0 to 100]
  Week 52: number analyzed (Participants) | 4
  Week 52 | 75.8 [40 to 100]

3. Secondary Outcome: Proportion of Patients Achieving mNAPSI of 0 in All Fingernails at Weeks 36 and 52.
Description: as for outcome 1
Time Frame: 36 and 52 weeks
Population: This was not measured.
Arm/Group | Study Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Percent Change in Patient Reported Nail Pain, as Based on the Nail Pain VAS Score, at Week 52 Compared to Baseline Score.
Description: Nail pain VAS is a subjective survey completed by patients. Scores range from 0 to 100 (0=no pain ; 100 = as severe pain as you can imagine). This outcome measure was completed by subtracting the value at Week 52 from the original value at baseline. This was a decrease, which was then divided by the baseline value and multiplied by 100.
Time Frame: 52 weeks
Population: Participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: percent change in nail pain score
Arm/Group | Study Group
Number analyzed (Participants) | 4
percent change in nail pain score | -50.42 (2.26)

5. Secondary Outcome: Pain Change in Psoriatic Arthritis (PsA) Symptoms at Week 52 Compared to Baseline, in Patients Who Self-identify as Having Psoriatic Arthritis at Baseline.
Description: Symptoms will be assessed using a visual analogue scale (VAS) for reporting psoriatic arthritis pain, which is a subjective survey that patients will complete on a scale of 0 to 100 (0= no pain ; 100 = as severe pain as you can imagine).This outcome measure was completed by subtracting the value at Week 52 from the original value at baseline. This was a decrease, which was then divided by the baseline value and multiplied by 100.
Time Frame: 52 weeks
Population: Participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage change in PsA pain symptoms
Arm/Group | Study Group
Number analyzed (Participants) | 4
percentage change in PsA pain symptoms | -28.97 (3.2)

6. Secondary Outcome: Safety Adverse Effects Will be Assessed at Each Visit
Description: Patients will be asked about illnesses and other health related events while taking part in the study.
Time Frame: 52 weeks
Population: All participants were asked about illnesses and other health related events during their time in the study. All were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 12
Participants
  Nausea | 5
  Abdominal pain | 1
  Acne | 1
  Acute gout | 2
  Acute eye vision loss | 1
  Bronchitis | 1
  Diarrhea | 1
  Emesis | 1
  Headache | 2
  Increased bowel movement | 1
  Psoriasis flare | 1
  Wrist skin infection | 1
  Salmonella | 1
  Upper respiratory infections | 3
  Viral Gastroenteritis | 1
  Worsened Asthma | 1
  Dyspepsia | 1
  Acute stroke | 1

7. Secondary Outcome: Proportion of Patients Achieving a mNAPSI 75 Response, as Defined by 75% or Greater Reduction Over Baseline in mNAPSI Score at Weeks 12, 24, 36, 48, and 52 for the Target Fingernail.
Description: as for outcome 2
Time Frame: 12, 24, 36, 48, and 52 weeks
Population: Data was not collected for this outcome.
Arm/Group | Study Group
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage Change From Baseline in mNAPSI.
Description: mNAPSI is an objective scoring system administered by trained health care providers. Scores range from 0 (no nail disease) to 130 (complete nail involvement in all ten nails.). For week 36 we averaged each participants mNAPSI percent change from baseline to week 36. We did the same thing for week 52
Time Frame: 36 and 52 weeks
Population: Participants were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: percent change
Units Other Than Participants: Nails
Arm/Group | Study Group
Number analyzed (Participants) | 6
Number analyzed (Nails) | 60
percent change
  Week 36 | 17.1 [10 to 60]
  Week 52: number analyzed (Participants) | 4
  Week 52 | 30 [10 to 62.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entirety of the study, 52 weeks for each participant
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=12)
Acute Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=12)
Nausea (General disorders) | 5 (7)
Abdominal Pain (General disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
acute gout (General disorders) | 2 (2)
Acute Eye Vision Loss (Eye disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diarrhea (General disorders) | 1 (1)
Emesis (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Increased Bowel Movements (General disorders) | 1 (1)
Psoriasis Flare (Skin and subcutaneous tissue disorders) | 1 (1)
Wrist Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Salmonella (General disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Viral Gastroenteritis (General disorders) | 1 (1)
Worsened Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03022617/Prot_SAP_000.pdf